CLINICAL TRIAL: NCT06721663
Title: Effect of Multisensory Environment Stimulation Therapy on Postural Control in Spastic Hemiplegic Cerebral Palsy
Brief Title: Multisensory Environment Stimulation Therapy on Postural Control in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Assistant Professor of Neurology and Neurosurgery Faculty of Physical Therapy October 6 University, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012005472
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental)
  Interventions: Other: Multisensory environment stimulation therapy; Other: selected physical therapy intervention
- control group (Experimental)
  Interventions: Other: selected physical therapy intervention

INTERVENTIONS:
Other: Multisensory environment stimulation therapy — A Multi Sensory Environment is a dedicated space or room where sensory stimulation can be controlled (intensified or reduced), presented in isolation or combination, packaged for active or passive interaction
  Arms: study group
Other: selected physical therapy intervention — therapeutic balance training and functional therapeutic exercises

SUMMARY:
To investigate the Effect of Multisensory environment stimulation therapy on postural control in spastic hemiplegic cerebral palsy.

DETAILED DESCRIPTION:
Fortypatients with spastic hemiplegic cerebral palsy will participate in this study.

The patients will randomly be divided into two equal groups; the control group which received the selected exercise program and the study group received the same exercise training program in addition to Multisensory environment stimulation therapy, three times per week for three months. The evaluation methods are BIODEX, The Pediatric Balance Scale, and multidirection reach test

ELIGIBILITY:
Inclusion Criteria:

* - Forty children with cerebral palsy,
* Age will range as (9:12) years old
* spastic hemiplegic cerebral palsy
* Normal body mass index standardmore than 50th and less than 85th for age and sex compared to standard Egyptian growth charts adopted by the Faculty of Medicine, Cairo University and National Research Centre.
* Gross motor function classification system: level I&II

Exclusion Criteria:

* • difficulty to communicate or to understand program instructions

  * any other neurological deficits or orthopaedic abnormalities,
  * secondary musculoskeletal complication
  * vestibular problems

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
biodex balance system | three months
  EVALUATION OF POSTURAL BALANCE USINGTHE BIODEX BALANCE SYSTEM
The Pediatric Balance Scale | three months
  used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.

SECONDARY OUTCOMES:
multidirection reach test | three months
  The Multi-Directional Reach Test (MDRT) measures balance and the limits of stability in the anterior-posterior and medial-lateral directions by testing how far an individual can voluntarily reach forward, to the right, to the left, and lean backward, while standing with their feet flat on the ground

CONTACTS AND LOCATIONS:
Locations (1):
- Lama S Mahmoud, Al Jīzah, Select State, Egypt